CLINICAL TRIAL: NCT02284893
Title: A 26-week International, Multicenter, Randomized, Double-Blind, Active Controlled, Parallel Group, Phase 3bTrial With a Blinded 26-week Long -Term Extension Period to Evaluate the Efficacy and Safety of Saxagliptin Co-administered With Dapagliflozin in Combination With Metformin Compared to Sitagliptin in Combination With Metformin in Adult Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control on Metformin Therapy Alone
Brief Title: Study to Evaluate the Efficacy and Safety of Saxagliptin Co-administered With Dapagliflozin in Combination With Metformin Compared to Sitagliptin in Combination With Metformin in Adult Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control on Metformin Therapy Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CV181-363; 2014-001102-17 (EudraCT Number)
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Results first posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; dapagliflozin; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A1:Saxagliptin / Placebo + Dapagliflozin / Placebo (Experimental): Saxagliptin 5 mg and matching placebo 0 mg (once daily) plus Dapagliflozin 10 mg and matching placebo 0 mg (once daily)
  Interventions: Drug: Saxagliptin; Drug: Dapagliflozin; Drug: Placebo matching with Saxagliptin; Drug: Placebo matching with Dapagliflozin
- A2: Sitagliptin / placebo (Experimental): Sitagliptin 100 mg and matching placebo 0 mg (once daily)
  Interventions: Drug: Sitagliptin; Drug: Placebo matching with Sitagliptin

INTERVENTIONS:
Drug: Saxagliptin — administered orally once daily
  Arms: A1:Saxagliptin / Placebo + Dapagliflozin / Placebo
Drug: Dapagliflozin — administered orally once daily
  Arms: A1:Saxagliptin / Placebo + Dapagliflozin / Placebo
Drug: Sitagliptin — administered orally once daily
  Arms: A2: Sitagliptin / placebo
Drug: Placebo matching with Saxagliptin — administered orally once daily
  Arms: A1:Saxagliptin / Placebo + Dapagliflozin / Placebo
Drug: Placebo matching with Dapagliflozin — administered orally once daily
  Arms: A1:Saxagliptin / Placebo + Dapagliflozin / Placebo
Drug: Placebo matching with Sitagliptin — administered orally once daily
  Arms: A2: Sitagliptin / placebo

SUMMARY:
Study will evaluate if a combination of saxagliptin and dapagliflozin added concurrently to metformin in combination with diet and exercise is superior to sitagliptin added to metformin in combination with diet and exercise in reducing mean HbA1c over a treatment period of 26 weeks.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Patients with Type 2 diabetes mellitus (T2DM) with inadequate glycemic control, defined as a central laboratory glycosylated hemoglobin (HbA1c) ≥8.0% and ≤ 10.5 % obtained at the screening visit
* Subjects should have been taking the same daily dose of metformin ≥ 1500 mg for at least 8 weeks prior to the enrollment visit and with no intake of other antihyperglycemic therapy for more than 14 days (consecutive or not) during 12 weeks prior to screening
* BMI > 20.0 kg/m2 at the enrollment visit
* Males and Females, age ≥18 years old at time of screening visit
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug
* Women must not be breastfeeding

Exclusion Criteria:

* Clinically diagnosed with Type I diabetes, known diagnosis of Maturity Onset Diabetes of Young (MODY), secondary diabetes mellitus or diabetes insipidus
* History of diabetic ketoacidosis
* Any of the following cardiovascular (CV)/Vascular Diseases within 3 months of the enrollment visit

  * Myocardial infarction
  * Cardiac surgery or revascularization (coronary artery bypass surgery Coronary Artery Bypass Graft [(CABG)]/percutaneous transluminal coronary angioplasty percutaneous transluminal coronary angioplasty [(PTCA)])
  * Unstable angina
  * Unstable congestive heart failure (CHF)
  * Transient ischemic attack (TIA) or significant cerebrovascular disease
  * Unstable or previously undiagnosed arrhythmia
  * Congestive heart failure, defined as New York Heart Association (NYHA) Class III and IV, unstable or acute congestive heart failure and/or known left ventricular ejection fraction of ≤ 40%
* Renal Disease
* Hepatic Diseases
* Hematological and Oncological Disease/Conditions
* Hemoglobin ≤ 11.0 g/dL (110 g/L) for men; hemoglobin ≤ 10.0 g/dL (100 g/L) for women
* Abnormal Free T4

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2014-09-09 (Actual); Primary Completion 2016-09-20 (Actual); Study Completion 2016-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Astra Zeneca, Study Director — AstraZeneca
Locations (70):
- United States (37):
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Huntington Beach, California
  - Research Site, Huntington Park, California
  - Research Site, Lomita, California
  - Research Site, Los Angeles, California
  - Research Site, Northridge, California
  - Research Site, Norwalk, California
  - Research Site, Paramount, California
  - Research Site, Sacramento, California
  - Research Site, Tarzana, California
  - Research Site, Tustin, California
  - Research Site, Golden, Colorado
  - Research Site, Coral Gables, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Council Bluffs, Iowa
  - Research Site, Crestview Hills, Kentucky
  - Research Site, Charlotte, North Carolina
  - Research Site, Morehead City, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Norman, Oklahoma
  - Research Site, Columbia, South Carolina
  - Research Site, Bristol, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, North Richland Hills, Texas
  - Research Site, Pasadena, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Manassas, Virginia
  - Research Site, Suffolk, Virginia
  - Research Site, Kenosha, Wisconsin
- Hungary (6):
  - Research Site, Baja
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Gyula
  - Research Site, Nyíregyháza
  - Research Site, Szekszárd
- Mexico (5):
  - Research Site, Aguascalientes
  - Research Site, Chihuahua City
  - Research Site, Cuautla
  - Research Site, Guadalajara
  - Research Site, Monterrey
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Opole
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Romania (8):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Buzău
  - Research Site, Craiova
  - Research Site, Galati
  - Research Site, Oradea
  - Research Site, Satu Mare
  - Research Site, Timișoara
- South Africa (7):
  - Research Site, Boksburg North
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, Lenasia
  - Research Site, Moloto South
  - Research Site, Soweto

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 461 Patients were Randomized into the study, 411 patients completed the 26 weeks part. Out of them 402 patients continued into the additional 26 week part. Out of them 378 patients completed the 52 weeks period (26+26 weeks).
Groups:
- SAXA + DAPA + MET: Saxagliptin 5-mg tablet+Dapagliflozin 10-mg tablet+Placebo capsules matching the sitagliptin 100-mg capsules+Metformin background therapy
- SITA + MET: Placebo tablet matching the saxagliptin 5-mg tablet +Placebo tablet matching the dapagliflozin 10-mg table+Sitagliptin 100-mg capsules +Metformin background therapy
Period: 26 Week (Short Term)
Arm/Group | SAXA + DAPA + MET | SITA + MET
Started | 232 | 229
Completed | 213 | 198
Not Completed | 19 | 31
Not completed — Adverse Event | 1 | 9
Not completed — Discontinuation by the subject | 2 | 2
Not completed — Withrawal of the consent by the subject | 7 | 10
Not completed — Lost to Follow-up | 3 | 1
Not completed — Subject no longer meets study criteria | 5 | 8
Not completed — Other | 1 | 1
Period: 52 Week (Long Term)
Arm/Group | SAXA + DAPA + MET | SITA + MET
Started | 209 | 193
Completed | 198 | 180
Not Completed | 11 | 13
Not completed — Adverse Event | 3 | 1
Not completed — Subject no longer meets study criteria | 0 | 1
Not completed — Withrawal of the consent by the subject | 4 | 6
Not completed — Lost to Follow-up | 2 | 2
Not completed — Non-Compliance | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SAXA + DAPA + MET | SITA + MET | Total
Number analyzed (Participants) | 232 | 229 | 461
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (8.87) | 55.8 (9.55) | 55.9 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 119 | 251
  Male | 100 | 110 | 210
Region of Enrollment [Number; unit: participants]
  Europe | 72 | 74 | 146
  North America | 114 | 113 | 227
  Central America | 46 | 42 | 88

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in HbA1c
Time Frame: Baseline (randomization) to Week 26
Population: The Randomized Subjects data set consists of all randomized subjects who received at least
  1 dose of double-blind study drug during the double-blind treatment period. Data in this data set were analyzed based on randomized treatment group, even if the treatment they received was different
Measure: Least Squares Mean (Standard Error); unit: percentage (%)
Groups:
- Saxagliptin + Dapagliflozin + Metformin Group: Saxagliptin 5-mg tablet +Dapagliflozin 10-mg tablet+Metformin background therapy +Placebo capsules matching the sitagliptin 100-mg capsules
Arm/Group | Saxagliptin + Dapagliflozin + Metformin Group | SITA + MET
Number analyzed (Participants) | 224 | 219
percentage (%) | -1.41 (0.0696) | -1.07 (0.0719)
Statistical Analysis 1: Comparison: Saxagliptin + Dapagliflozin + Metformin Group vs SITA + MET; Test type: Superiority; p = 0.0008, Mixed Models Analysis; Mean Difference (Final Values) = -0.34, Standard Error of Mean 0.1001

2. Secondary Outcome: Percent of Subjects Achieving a Therapeutic Glycemic Response, Defined as HbA1c < 7.0%
Time Frame: week 26
Population: randomized subjects
Measure: Number; unit: Percentage of subjects
Arm/Group | Saxagliptin + Dapagliflozin + Metformin Group | SITA + MET
Number analyzed (Participants) | 224 | 219
Percentage of subjects | 37.3 (3.150) | 25.1 (2.871)
Statistical Analysis 1: Comparison: Saxagliptin + Dapagliflozin + Metformin Group vs SITA + MET; Test type: Superiority; p = 0.0034, Regression, Logistic; the analysis was by Zhang et.al. method with adjustment for baseline A1c.The measure of interest is NOT odds ratio but Risk Difference; Risk Difference (RD) = 12.2, Standard Error of Mean 4.175

3. Secondary Outcome: Mean Change in Total Body Weight
Time Frame: Baseline (randomization) to Week 26
Population: randomized subjects
Measure: Mean (Standard Error); unit: kg
Arm/Group | Saxagliptin + Dapagliflozin + Metformin Group | SITA + MET
Number analyzed (Participants) | 224 | 219
kg | -1.86 (0.2010) | -0.51 (0.2078)
Statistical Analysis 1: Comparison: Saxagliptin + Dapagliflozin + Metformin Group vs SITA + MET; Test type: Superiority; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -1.35, Standard Error of Mean 0.2891

4. Secondary Outcome: Mean Change in Fasting Plasma Glucose (FPG)
Time Frame: Baseline (randomization) to Week 26
Population: randomized subjects
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Saxagliptin + Dapagliflozin + Metformin Group | SITA + MET
Number analyzed (Participants) | 224 | 219
mg/dl | -31.9 (2.538) | -11.0 (2.668)
Statistical Analysis 1: Comparison: Saxagliptin + Dapagliflozin + Metformin Group vs SITA + MET; Test type: Superiority; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -20.9, Standard Error of Mean 3.682

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: Including Data After Rescue, Treated Subjects
Groups:
- Sita + Met: Placebo tablet matching the saxagliptin 5-mg tablet+Placebo tablet matching the dapagliflozin 10-mg tablet+Sitagliptin 100-mg capsules+Metformin background therapy
Arm/Group | SAXA + DAPA + MET | Sita + Met
All-Cause Mortality (participants affected / at risk) | 0/232 | 0/229
Serious Adverse Events (participants affected / at risk) | 9/232 | 13/229
Other Adverse Events (participants affected / at risk) | 112/232 | 123/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAXA + DAPA + MET (N=232) | Sita + Met (N=229)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0
PALPITATIONS (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 0 | 1
MITRAL VALVE PROLAPSE (Cardiac disorders) | 0 | 1
TACHYCARDIA (Cardiac disorders) | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
ANAL FISSURE (Gastrointestinal disorders) | 0 | 1
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
POST LAMINECTOMY SYNDROME (Injury, poisoning and procedural complications) | 1 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 1
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
DYSFUNCTIONAL UTERINE BLEEDING (Reproductive system and breast disorders) | 1 | 0
ENDOMETRIOSIS (Reproductive system and breast disorders) | 0 | 2
LUMBAR RADICULOPATHY (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 2
SEPSIS (Infections and infestations) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 2
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SAXA + DAPA + MET (N=232) | Sita + Met (N=229)
NASOPHARYNGITIS (Infections and infestations) | 18 | 12
HEADACHE (Nervous system disorders) | 13 | 10
URINARY TRACT INFECTION (Renal and urinary disorders) | 10 | 7
INFLUENZA (Infections and infestations) | 8 | 11
BRONCHITIS (Infections and infestations) | 8 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 | 8
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 9
DYSLIPIDAEMIA (Congenital, familial and genetic disorders) | 5 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 | 2
SINUSITIS (Infections and infestations) | 5 | 2
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 5 | 2
GASTROENTERITIS (Infections and infestations) | 4 | 5
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 5 | 1
HYPERTENSION (Vascular disorders) | 3 | 8
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 7
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 6
DIARRHOEA (Gastrointestinal disorders) | 2 | 6
ANAEMIA (Blood and lymphatic system disorders) | 1 | 7
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 5
GASTRITIS (Gastrointestinal disorders) | 1 | 5
HYPERGLYCAEMIA (Endocrine disorders) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI to provide AstraZeneca (AZ) with an opportunity to review/comment on drafts of publication and review final draft at least 30 days in advance of submission for publication or public presentation (15 days for an abstract or poster). If requested agree to delay submission or presentation for an additional period, not more than additional 90 days, to allow AZ to file a patent or application to preserve our rights in any intellectual property disclosed in the publication.